CLINICAL TRIAL: NCT06085716
Title: Combination Therapy for Cancer Related Fatigue in Patients With Metastatic Cancers
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-0466; NCI-2023-08682 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Cancers; Fatigue
MeSH Terms: conditions — Neoplasms; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Psychoeducational Intervention (Experimental): Participants will be randomly assigned to 1 of 3 study groups. The study treatment participants get will be chosen by chance, like rolling the dice. Both participants and the study staff will know which treatment you were assigned:
  Interventions: Behavioral: Psychoeducational Intervention
- Open Label Placebo (Experimental): Participants will be randomly assigned to 1 of 3 study groups. The study treatment participants get will be chosen by chance, like rolling the dice. Both participants and the study staff will know which treatment you were assigned:
  Interventions: Drug: Open Label Placebo
- Psychoeducational Intervention+Placebo (Experimental): Participants will be randomly assigned to 1 of 3 study groups. The study treatment participants get will be chosen by chance, like rolling the dice. Both participants and the study staff will know which treatment you were assigned:
  Interventions: Behavioral: Psychoeducational Intervention+Placebo

INTERVENTIONS:
Behavioral: Psychoeducational Intervention — Participants in the PI group will complete the educational sessions only.
  Arms: Psychoeducational Intervention
Drug: Open Label Placebo — This group will only take placebo capsules every day.
  Arms: Open Label Placebo
Behavioral: Psychoeducational Intervention+Placebo — This group will take the placebo capsules every day, as well as completing the educational sessions.
  Arms: Psychoeducational Intervention+Placebo

SUMMARY:
To find out if combining psychoeducational interventions (such as education, counseling, and self-managed therapies) with an open-label placebo can help to improve your quality of life better than either the psychoeducational interventions or the placebo alone.

DETAILED DESCRIPTION:
Primary Objectives:

1. To determine if the combination therapy of PI with OLP (combination therapy group) is superior to PI alone group in the treatment of cancer-related fatigue (CRF) as measured by the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) scale.

We hypothesize that the combination of OLP+PI in these patients will result in a greater reduction of CRF compared to PI alone.

Secondary Objectives:

1. To determine if Combination Therapy group is superior to PI Only group for the treatment of CRF at 3 months and 6 months after treatment. We hypothesize that the combination of OLP+PI in these patients will result in a greater reduction of CRF after 3 months and 6 months after treatment

3. To determine the effects of combination therapy on fatigue-related quality-of-life, mood, sleep-wake activity, cognitive measures, and inflammation. We will assess measures including quality of life (Functional Assessment of Cancer Therapy - General, FACT- G), multidimensional fatigue (Multidimensional Fatigue Symptom Inventory, MFSI-SF), sleep disturbance (PROMIS-sleep), anxiety (Hospital Anxiety and Depression Scale - HADS), depressed mood (HADS), cognitive function (Symbol digit modality test, SDMT), sleep/wake time activity (actigraphy), and inflammation (C-reactive protein levels).

We hypothesize that combination therapy will result in improvements in CRF-related quality of life, mood, sleep-wake activity, and cognitive measures.

ELIGIBILITY:
Inclusion Criteria:

1. Be advanced cancer patients (incurable metastatic), having fatigue with severity of 4/10, on a 0-10 scale (Edmonton Symptom Assessment Scale) for at least 2 weeks.
2. Have no clinical evidence of cognitive failure as evidenced by treating clinician assessment at screening (Memorial Delirium Assessment Scale of less than 13/30).
3. Be aged 18 years or older.
4. Be willing to complete in-person or with research staff, and able to complete Psychoeducational intervention either in person or virtually within Texas.
5. Have a hemoglobin level of ≥10 g/dL within 2 weeks of enrollment.
6. Be able to understand the description of the study and sign a written informed consent.
7. Have a ECOG performance status score of 0 to 2; and
8. Be seen at an outpatient clinic at MD Anderson Cancer Center's (MDA) main campus or its Houston Area Locations (HALs)

Exclusion Criteria:

1. Have a major contraindication to placebo (e.g., allergy or hypersensitivity to study medications or their constituents), or conditions making adherence difficult as determined by the attending physician.
2. Be unable to complete the baseline assessment forms or to understand the recommendations for participation in the study.
3. Be pregnant or become pregnant while on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Centerr, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org